CLINICAL TRIAL: NCT01395446
Title: The Application of an Electronic Nose in the Early Detection of ASpergillosis
Brief Title: Application of an Electronic Nose in the Early Detection of ASpergillosis
Acronym: AENEAS
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, K. de Heer, Drs. K. de Heer, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 28062009
Record Dates: First submitted 2011-06-29; First posted 2011-07-15 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Pulmonary Invasive Aspergillosis
MeSH Terms: conditions — Invasive Pulmonary Aspergillosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — BAL
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- prolonged neutropenic patients: patients that will undergo treatment for a hematological malignancy expected to result in grade 4 neutropenia of prolonged duration

SUMMARY:
The purpose of this study is to establish the accuracy with which the eNose can discriminate patients with invasive pulmonary aspergillosis from controls.

ELIGIBILITY:
Inclusion Criteria:

Patients that

1. are 18 years of age or older
2. will undergo treatment for a hematological malignancy expected to result in grade 4 neutropenia (according to CTCAE 3.0, i.e. <0.5 x 109 neutrophils/L) of prolonged duration (i.e., more than 7 days), e.g. hematopoietic stem cell transplantation or induction/consolidation treatment for acute myeloid leukaemia
3. have given written informed consent

Exclusion Criteria:

1. a previously diagnosed invasive mycosis
2. the inability to perform the breathing manoeuvre needed for eNose-analysis of exhaled air

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients that will undergo treatment for a hematological malignancy expected to result in grade 4 neutropenia of prolonged duration
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2010-01; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
accuracy with which the Cyranose can discriminate between patients with probable or proven invasive pulmonary aspergillosis and neutropenic controls with fever | 4 days
  The cross-validated accuracy with which the Cyranose can discriminate between patients with probable or proven invasive pulmonary aspergillosis and neutropenic controls with fever, defined as the percentage of correctly classified patients using the leave-one out method

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hematology, Academic Medical Center, Amsterdam, Netherlands